CLINICAL TRIAL: NCT00635583
Title: Influence of Dairy on Bone Accrual and Bone Size and Fat and Lean Mass in Early Pubertal Overweight vs. Healthy-weight Boys and Girls
Brief Title: The Effect of Dairy on Bone Mass and Body Composition in 4th-8th Grade Boys and Girls
Acronym: B3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Indiana University School of Medicine (Other); Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1482
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Bone; Dairy Intervention; Girls; Boys; Calcium; Bone Mineralization; Peak Bone Mass; Bone and Bones; Female; Male; Adolescent; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Increased Dairy Consumption (Experimental): Increased Dairy Consumption - Each subject in this arm will receive three additional servings of dairy to consume each day for 18 months.
  Interventions: Other: Increased Dairy Consumption
- Control (No Intervention): This group will not receive the intervention but will continue their normal diet; they will act as the control.

INTERVENTIONS:
Other: Increased Dairy Consumption — 3 additional servings of dairy (two of which must be milk or yogurt)
  * 8 oz milk
  * 6 oz yogurt
  * 1.5 oz cheese
  Other Names: Prairie Farms Milk; Prairie Farms Yogurt
  Arms: Increased Dairy Consumption

SUMMARY:
Building stronger bones during pubertal growth could reduce lifelong fracture risk. This project is an 18 month dairy intervention study for overweight and healthy weight 4th-8th grade boys and girls. Half of the girls will receive dairy products to add to their habitual diet (milk, yogurt, and cheese) to equal three products per day, while the other half will remain on their normal diet. All participants will attend four study visits, each 6 months apart. At these visits height, weight, bone density and geometry, and fat and lean mass will be measured. This study aims to show that meeting calcium requirements by eating dairy products builds bigger, stronger bones, and that this effect may be enhanced in overweight boys and girls. The effect of the dairy intervention on body fat, lean mass, and weight, as well as the mechanisms and predictors of changes in bone mass and size and body composition will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Males and females in 4th-8th grade
* Generally healthy
* BMI percentile 5-70% for age or >85% for age
* Baseline calcium intake less than or equal to 800mg/d

Exclusion Criteria:

* History of any illness known to affect bone mass accrual (diabetes, inflammatory bowel disease, childhood malignancy).
* A broken bone in the last six months.
* Consume more than 800 mg Calcium/d.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Changes in bone density and geometry as measured with DEXA and pQCT. | 18 months

SECONDARY OUTCOMES:
Changes in fat and lean body mass as measured with DEXA. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Purdue University
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Purdue University, West Lafayette, Indiana

REFERENCES:
- [Derived] Vogel KA, Martin BR, McCabe LD, Peacock M, Warden SJ, McCabe GP, Weaver CM. The effect of dairy intake on bone mass and body composition in early pubertal girls and boys: a randomized controlled trial. Am J Clin Nutr. 2017 May;105(5):1214-1229. doi: 10.3945/ajcn.116.140418. Epub 2017 Mar 22. PMID 28330908